CLINICAL TRIAL: NCT02221622
Title: Allopregnanolone Regenerative Therapeutic for MCI/AD: Dose Finding Phase 1
Brief Title: Allopregnanolone for Mild Cognitive Impairment Due to Alzheimer's Disease or Mild AD
Acronym: Allo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AlloPhase1; 1UF1AG046148 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-08-20 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Alzheimer's disease; Mild Cognitive Impairment; Dementia; Regenerative therapeutic
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Pregnanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Allopregnanolone 2 mg (Experimental): Drug: Allopregnanolone injection (intravenous solution) once per week for 12 weeks
  Interventions: Drug: Allopregnanolone injection (intravenous solution)
- Allopregnanolone 4 mg (Experimental): Drug: Allopregnanolone injection (intravenous solution) once per week for 12 weeks
  Interventions: Drug: Allopregnanolone injection (intravenous solution)
- Allopregnanolone 6-18 mg (Experimental): Drug: Allopregnanolone injection (intravenous solution) once per week for 12 weeks
  Interventions: Drug: Allopregnanolone injection (intravenous solution)
- Placebo (Placebo Comparator): Drug: Placebo injection (intravenous solution) once per week for 12 weeks
  Interventions: Drug: Placebo injection (intravenous solution)

INTERVENTIONS:
Drug: Allopregnanolone injection (intravenous solution) — Allopregnanolone intravenous infusion
  Other Names: 3α,5α-tetrahydroprogesterone; 3α-hydroxy-5α-pregnan-20-one
  Arms: Allopregnanolone 2 mg; Allopregnanolone 4 mg; Allopregnanolone 6-18 mg
Drug: Placebo injection (intravenous solution) — Placebo intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of allopregnanolone, a naturally occurring brain steroid, in mild cognitive impairment and early Alzheimer's disease participants. The primary goal is to determine the maximally tolerated dose.

DETAILED DESCRIPTION:
1) Each dose group will be comprised of 8 participants (6 randomized to allopregnanolone; 2 randomized to placebo) administered one dose of allopregnanolone or placebo once per week for 12 weeks. A higher dose will be administered to the next group of participants when the lower dose is shown to be safe and tolerable. 2) Pharmacokinetic analyses will be conducted on blood samples taken from participants at the beginning and end of the trial. 3) The trial will assess safety including via MRI brain imaging.

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal women
* 55 years of age or older
* Diagnosis of MCI due to AD or mild AD
* MMSE > 20 at screen
* Capacity to provide informed consent
* Residing in the community with a caregiver able to accompany the patient to clinic visits
* No medical contraindications to participation
* Willingness to comply with study procedures

Exclusion Criteria:

* Use of benzodiazepines, sedative/hypnotics, anticonvulsants, antipsychotics, and other drugs that might interact with the GABA-A receptor complex
* Seizure disorder, history of stroke, focal brain lesion, traumatic brain injury, substance abuse, malignancy
* Clinically significant laboratory or ECG abnormality
* MRI indicative of any other significant abnormality, including but not limited to evidence of a cerebral contusion, encephalomalacia, aneurysms, vascular malformations, subdural hematoma, or space occupying lesions
* Any condition that would contraindicate an MRI such as the presence of metallic objects in the eyes, skin, heart, or body

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Safety profile: Adverse events | From Baseline to week 16
  Incidence and severity of treatment emergent adverse events assessed weekly per treatment arm.
Safety profile: Clinical laboratory measurements | From Baseline to week 13
  Evaluating the proportion of subjects exceeding pre-established critical values per treatment arm:
  Alanine aminotransferase (ALT, U/L) > 5 times upper normal limit Aspartate aminotransferase (AST, U/L) > 5 times upper normal limit Total serum bilirubin (mg/dl) > 2 times upper normal limit Serum creatinine (mg/dl) > 2 times upper normal limit Serum creatine phosphokinase (U/L) > 5 times upper normal limit
Safety profile: ARIA | From Baseline to week 13
  MRI based assessment of amyloid related imaging abnormalities (ARIA); proportion of subjects with ARIA
Safety profile: Physical and neurological examination | From Baseline to week 16
  To evaluate the proportion of abnormal examination findings of subjects in each treatment arm.
Tolerability - Maximum tolerated dose (MTD) | From Baseline to week 12
  Onset of sedation will define the upper most limit of drug dose

SECONDARY OUTCOMES:
Pharmacokinetic profile after single and multiple doses: Maximum Concentration (Cmax) | Weeks: 1 and 12
  Measurement of maximum concentration
Pharmacokinetic profile after single and multiple doses: time attain to Cmax (Tmax) | Weeks: 1 and 12
  Time to attain maximum concentration.
Pharmacokinetic profile after single and multiple doses: Area under the curve (AUC) | Weeks: 1 and 12
  Pharmacokinetic parameter.
Pharmacokinetic profile after single and multiple doses: Drug Clearance (CL) | Weeks: 1 and 12
  Pharmacokinetic parameter.
Pharmacokinetic profile after single and multiple doses: apparent volume of distribution at steady state (Vss) | Weeks: 1 and 12
  Pharmacokinetic parameter.
Cognitive tests (ADAS-Cog; MMSE/MoCA; ADCS-CGIC; CogState) | Baseline to Week 13
  Alzheimer's disease Assessment Scale Cognitive Subscale 14 (ADAS-Cog); Mini-Mental State Exam (MMSE); Montreal Cognitive Assessment (MoCA); Alzheimer's disease Cooperative Study Clinical Global Impression of Change (ADCS-CGIC); CogState 12-min battery (CogState)
Brain MRI volumetrics | Baseline and Week 13
  Gray matter, white matter and hippocampal volume measurements, including subfield analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta D Brinton, Ph.D., Principal Investigator — University of Southern California; Lon S Schneider, M.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California - Alzheimer Disease Research Center - Healthcare Consultation Center II, Los Angeles, California, United States

REFERENCES:
- [Derived] Hernandez GD, Solinsky CM, Mack WJ, Kono N, Rodgers KE, Wu CY, Mollo AR, Lopez CM, Pawluczyk S, Bauer G, Matthews D, Shi Y, Law M, Rogawski MA, Schneider LS, Brinton RD. Safety, tolerability, and pharmacokinetics of allopregnanolone as a regenerative therapeutic for Alzheimer's disease: A single and multiple ascending dose phase 1b/2a clinical trial. Alzheimers Dement (N Y). 2020 Dec 16;6(1):e12107. doi: 10.1002/trc2.12107. eCollection 2020. PMID 33344752